CLINICAL TRIAL: NCT06778239
Title: Natural History Study to Determine Childhood-Onset Essential Hypertension Etiology
Brief Title: Childhood-Onset Essential Hypertension Natural History Study
Status: Recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001987; 001987-HG
Record Dates: First submitted 2025-01-15; First posted 2025-01-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-26

CONDITIONS: Hypertension; Essential Hypertension
Keywords: Blood Pressure; Pediatric; childhood hypertension; ESSENTIAL HYPERTENSION; Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected: Study participants that are 2-17 years old and have COEH or participants that are 18+ years old that were diagnosed with COEH when they were children.
- Unaffected: Study participants that are 2+ years old and have never been diagnosed with COEH.

SUMMARY:
Background:

Childhood-onset essential hypertension (COEH) is high blood pressure that develops in children and teens. High blood pressure is a major risk factor for heart disease. COEH is more likely to be caused by changes in genes rather than by factors like stress or diet. Researchers want to learn more about how changes in genes relate to COEH. They hope to use that information to develop better treatments for children with high blood pressure.

Objective:

This natural history study will look for genes and gene changes that may lead to COEH.

Eligibility:

People aged 2 years and older with COEH or who had COEH when they were children. Healthy relatives of those with COEH are also needed.

Design:

Participants will have one clinic visit per year for up to 10 years. All participants will have a physical exam. They will provide samples of blood and urine. At their first visit, they will have a swab (like a Q-tip) rubbed between their gums and cheeks. They may agree to having a skin biopsy; a piece of skin about the size of a pencil eraser will be removed.

Affected participants aged 2 to 17 years old will have additional tests:

* They will have sensors placed on their skin to look at their blood vessels and see how blood is moving in their bodies.
* They will lie or stand while a machine measures the amount of fat and muscle in their bodies.
* They will have an ultrasound; a wand will be rubbed against their skin to take pictures of their kidneys.

Other things are optional for all participants:

* They may have photographs taken of their bodies.
* They may have tests of their heart function.
* They may have different types of imaging scans.

DETAILED DESCRIPTION:
Study Description:

This study seeks to identify molecular processes and genetics that contribute to the development of childhood-onset essential hypertension (COEH) in a diverse cohort of children. Identification of blood pressure (BP)-regulating pathway(s) involved in COEH will allow for targeted and individualized therapy.

Objectives:

Primary Objective:

Elucidate the molecular genetic processes associated with developing COEH.

Secondary Objective:

Characterize the vascular, clinical, and laboratory phenotypes seen in patients with COEH.

Endpoints:

Primary Endpoint:

Evidence that saturation of the allelic spectrum for COEH has been reached.

Secondary Endpoint:

Completion of exhaustive phenotyping on COEH patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an affected individual must meet one of the following criteria:

* Age 2-12 years at time of enrollment with a BP of at least >95th percentile or 120/80 mm Hg verified via medical record review and a willingness to provide biological samples, undergo physical exam, provide information related to family and medical history, and undergo imaging/body measurements (e.g., renal ultrasound)
* Age 13-17 years at time of enrollment with a BP of at least 130/80 mm Hg verified via medical record review and a willingness to provide biological samples, undergo physical exam, provide information related to family and medical history, and undergo imaging/body measurements (e.g., renal ultrasound)
* Age 18 years or more at time of enrollment with a medical history of meeting the criteria outlined in affected individual inclusion criteria 1 or 2, depending on age at diagnosis (verified via medical record review) and a willingness to provide biological samples, undergo physical exam, and provide information related to family and medical history

To be eligible to participate in this study, an unaffected individual must meet all of the following criteria:

* First-degree relative to a proband (first identified affected family member) in the study
* Willingness to provide biological samples, undergo physical exam, and provide information related to family and medical history

To be eligible to participate in this study, an individual with a candidate variant (regardless of known COEH status) must meet all of the following criteria:

* History of clinical and/or research genomic interrogation
* Positive genomic interrogation test result for candidate variant identified in earlier stages of study or in prior studies performed by study team
* Willingness to provide information related to family and medical history, provide access to relevant medical records, undergo physical exam, and undergo imaging/body measurements (if 2-17 years of age and evidence of COEH exists)

EXCLUSION CRITERIA:

An affected individual who meets any of the following criteria will be excluded from participation in this study:

* BMI >95th percentile
* Evidence that hypertension is secondary to a known condition (e.g., chronic kidney disease, aortopathy, sleep apnea, etc.)
* Impaired decision-making capability, with or without a legally-authorized representative

An unaffected individual who meets any of the following criteria will be excluded from participation in this study:

* Prior or current diagnosis of COEH
* Second-degree or greater relationship to proband
* Impaired decision-making capability, with or without a legally-authorized representative

An individual with a candidate variant (regardless of known COEH status) who meets any of the following criteria will be excluded from participation in this study:

* No prior genomic interrogation findings available for the study team to review to confirm positive candidate variant status
* Impaired decision-making capability, with or without a legally-authorized representative

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will come from hypertension, cardiology, nephrology (kidney), and pediatrician clinics. Participants can also sign themselves up for the study without being referred by their doctor.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2034-12-09 (Estimated); Study Completion 2034-12-09 (Estimated)

PRIMARY OUTCOMES:
Find all genes that cause COEH. | 10 years

SECONDARY OUTCOMES:
Identify all of the ways that COEH affects the body. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Hanchard, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001987-HG.html